CLINICAL TRIAL: NCT05446844
Title: Impact of Implementing a Nurse Caring Behavior Protocol on Postoperative Cardiac Patient Satisfaction: A Randomized Controlled Trial
Brief Title: A Nurse Caring Behavior Protocol on Postoperative Cardiac Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Suad Elsaman, Assistant professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Patient satisfaction
Record Dates: First submitted 2022-06-22; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Nurse-Patient Relations; Patient Satisfaction; Caring
Keywords: Cardiac patient; Nurse caring behaviors; Satisfaction
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A protocol group (Experimental): A protocol group received a nurse caring behavior protocol by the researcher
  Interventions: Other: A nurse caring behavior protocol
- A control group (Active Comparator): A control group received routine nursing care by the staff nurse
  Interventions: Other: Routine nursing care

INTERVENTIONS:
Other: A nurse caring behavior protocol — Nursing interventions based on caring behaviors protocol was provided as follows:
  * Caring behaviors during ICU admission and orientation processes included orienting patients to time, place, and person.
  * Caring behaviors during physical care informing patients regarding the purpose and expected duration of mechanical ventilator use.
  * Caring behaviors during psychological care included offering religious sound meditation.
  * Caring behaviors during social interaction included maintaining eye contact during nurse-patient interaction.
  * Caring behaviors during health teaching included providing health teaching for patients.
  * Caring behaviors during maintaining a safe healing environment included providing patients with an explanation regarding nursing activities.
  Arms: A protocol group
Other: Routine nursing care — Routine nursing care was concentrated mainly on hard skills of physically demanding care such as monitoring vital signs.
  Arms: A control group

SUMMARY:
the study aimed to evaluate the impact of implementing a nurse caring behavior (NCB) protocol on postoperative cardiac patient satisfaction.

DETAILED DESCRIPTION:
Critical care nurses need to comply with caring behaviors when caring for postoperative cardiac patients. Furthermore, patient satisfaction is a key indicator of nursing care quality. As such, this study focused on these critical issues considering the limited research available on the impact of caring behaviors on postoperative cardiac patient satisfaction. The study aimed to evaluate the impact of implementing a nurse caring behavior protocol on postoperative cardiac patient satisfaction. The study was conducted at a cardiac surgery intensive care unit of Alexandria Main University Hospital, Egypt. Sixty adults, conscious cardiac surgery patients, were included during the first 2 days following surgery. Patients were randomly assigned to either a control group, which received routine nursing care, or a protocol group, which received nursing care based on nurse care behaviors protocol through a simple randomization method. One tool was used "Postoperative Cardiac Patient Satisfaction with Nurse Caring Behaviors Evaluation Questionnaire". At the end of the second day, patients were asked regarding their satisfaction with the nursing care received based on caring behaviors. These nursing care included intensive care unit admission and orientation processes, physical care, psychological care, and social interaction between patient and nurse, providing health teaching, and maintaining a safe healing environment.

ELIGIBILITY:
Inclusion Criteria:

* Underwent cardiac surgery.

Exclusion Criteria:

* Unstable hemodynamics (systolic blood pressure less than 90).
* Uncontrolled dysrhythmias.
* Hemorrhage.
* Uncontrolled diabetes mellitus.
* Chronic respiratory diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with Intensive care unit admission and orientation processes based on caring behaviors questionnaire: | At the end of the second postoperative day
  The questionnaire includes statement items on nursing interventions based on nurse caring behaviors related to admission and orientation process such as (Nurses welcoming and identify themselves to the patients, Orientation provided by the nurse regarding time, place, and person and Orientation provided by the nurse regarding nursing activities that will be done). Each statement item was rated on a dichotomous scale of (satisfied, dissatisfied) after the researcher asked the patients to report whether they were satisfied with the care provided. Each statement item was scored as follows: satisfied = 1 and dissatisfied = 0.
Patient satisfaction with physical care based on caring behaviors questionnaire: | At the end of the second postoperative day
  The questionnaire includes statement items on nursing interventions based on nurse caring behaviors related to physical care which was provided to the patients such as (The manner at which nurses talk to patients, The ability of nurses to establish realistic goals, Responding to patient complaints, Nurse's helpfulness Nurses' availability, Praising the patients for performing activities). Each statement item was rated on a dichotomous scale of (satisfied, dissatisfied) after the researcher asked the patients to report whether they were satisfied with the care provided. Each statement item was scored as follows: satisfied = 1 and dissatisfied = 0.
Patient satisfaction with psychological care based on caring behaviors questionnaire. | At the end of the second postoperative day
  The questionnaire includes statement items on nursing interventions based on nurse caring behaviors related to psychological care which was provided to the patients such as (Dealing with patients and providing enthusiasm, Level of confidentiality that nurses provided to patients, Always repeating statements that instilled hope). Each statement item was rated on a dichotomous scale of (satisfied, dissatisfied) after the researcher asked the patients to report whether they were satisfied with the care provided. Each statement item was scored as follows: satisfied = 1 and dissatisfied = 0.
Patient satisfaction with social interaction based on caring behaviors questionnaire. | At the end of the second postoperative day
  The questionnaire includes statement items on nursing interventions based on nurse caring behaviors related to social interaction between patient and nurse such as (Duration of time nurses' spent with patients, Maintaining a cheerful disposition, Making patients feel at home, Nurse's ability to provide verbal reassurance, Nurse's ability to use the eye-to-eye contact with the patient). Each statement item was rated on a dichotomous scale of (satisfied, dissatisfied) after the researcher asked the patients to report whether they were satisfied with the care provided. Each statement item was scored as follows: satisfied = 1 and dissatisfied = 0.
Patient satisfaction with health teaching based on caring behaviors questionnaire. | At the end of the second postoperative day
  The questionnaire includes statement items on nursing interventions based on nurse caring behaviors related to health teaching which was provided to the patients such as (Information provided by the nurse regarding diagnosis, your rights, and treatment plan, Information provided by the nurse regarding postoperative activity, Information provided by the nurse regarding diagnostic procedures, Feasibility and clearness of the information provided by the nurse, Time at which the nurse provided information was enough and suitable for the patient). Each statement item was rated on a dichotomous scale of (satisfied, dissatisfied) after the researcher asked the patients to report whether they were satisfied with the care provided. Each statement item was scored as follows: satisfied = 1 and dissatisfied = 0.
Patient satisfaction with maintaining a safe healing environment based on caring behaviors questionnaire | At the end of the second postoperative day
  The questionnaire includes statement items on nursing interventions based on nurse caring behaviors related to maintaining a safe healing environment such as (Availability of comfort measures, such as lighting, noise control, and adequate blankets, Cleanliness and ventilation of the intensive care unit, Adequacy of sleeping time, Keeping patients away from unpleasant scenes, Availability glasses, hearing aids, and familiar objects). Each statement item was rated on a dichotomous scale of (satisfied, dissatisfied) after the researcher asked the patients to report whether they were satisfied with the care provided. Each statement item was scored as follows: satisfied = 1 and dissatisfied = 0.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandria University, Study Chair — Faculty of Nursing, Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickey PL, Angus PW, McLean AJ, Morgan DJ. Oxygen supplementation restores theophylline clearance to normal in cirrhotic rats. Gastroenterology. 1995 May;108(5):1504-9. doi: 10.1016/0016-5085(95)90700-9. PMID 7729643
- [Background] Salimi S, Tarbiat S. Predictors and priority of caring behaviours in intensive care units. Nurs Crit Care. 2021 Nov;26(6):523-530. doi: 10.1111/nicc.12590. Epub 2021 Jan 25. PMID 33496010
- [Background] Karabey T. Reflection of nurses' moral intelligence levels on care behaviors. Perspect Psychiatr Care. 2022 Oct;58(4):1622-1631. doi: 10.1111/ppc.12970. Epub 2021 Nov 24. PMID 34820855